CLINICAL TRIAL: NCT00564499
Title: A Scientific Research Program to Evaluate the Efficacy of SYMBICORT® 320/9μg in the Treatment of COPD in Real Life Environment by General Practitioners
Brief Title: SYMBICORT® in the Treatment of COPD
Acronym: SRP COPD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: SRP-RB-COPD-2005/1
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: COPD
Keywords: COPD; Symbicort; General Practitioners
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A Scientific Research Program to evaluate the efficacy of SYMBICORT® 320/9μg in the treatment of COPD in real life environment by General Practitioners

ELIGIBILITY:
Inclusion Criteria:

* patients (m/f) with COPD (GOLD stadium III and IV)

Exclusion Criteria:

* patients who recently quit smoking (<3months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Dates: Start 2006-03; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Louis, PR, Principal Investigator — Université Libre de Liège